CLINICAL TRIAL: NCT02615158
Title: Toddler Overweight Prevention: Comparison of Maternal and Toddler Intervention
Brief Title: Toddler Overweight Prevention Study Among Low-Income Families
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Johns Hopkins University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-27980; R01HD056099 (NIH); R03HD077156 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2015-11-26 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Overweight; Obesity; Depression
Keywords: Feeding practices; Diet; Physical activity; Prevention
MeSH Terms: conditions — Overweight; Obesity; Depression; Motor Activity | interventions — Nutritional Status; Psychological Tests; Child Restraint Systems

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Maternal Physical Activity and Nutrition (Experimental): A maternal intervention focusing on healthy diet and physical activity patterns for mothers.
  Interventions: Behavioral: Maternal Physical Activity and Nutrition
- Parenting (Experimental): A toddler parenting intervention focusing on parenting, limit setting, and development strategies.
  Interventions: Behavioral: Parenting
- Child Safety (Experimental): Attention control group. The parents received intervention to promote safety among toddlers.
  Interventions: Behavioral: Child Safety

INTERVENTIONS:
Behavioral: Maternal Physical Activity and Nutrition — At each session, mothers will identify a dietary goal for the next session (e.g., reduce soda intake). They will learn to track and evaluate their progress, setting new goals or modifying existing ones as necessary. Mothers will be given pedometers and shown how to keep a pedometer tracking chart. As with dietary choice, our objective is to have the mothers identify personal goals and strategies to achieve those goals, so they are more likely to continue to engage in physical activity after the intervention ends.
  Arms: Maternal Physical Activity and Nutrition
Behavioral: Parenting — Behavior and Development Related to Diet and Physical Activity. The toddler parenting intervention will include modules on toddler behavior and development. We will devote sessions to topics involving parenting toddlers, limit setting, and child development.
  Arms: Parenting
Behavioral: Child Safety — The intervention will focus on child safety issues, including car seat safety, fire safety, fall prevention, and poison prevention. Participants will set weekly child safety goals.
  Arms: Child Safety

SUMMARY:
The hypothesis is that toddlers with parents who are randomized to a parenting intervention and toddlers with parents who are randomized to the maternal intervention focused on maternal diet and physical activity will be more likely to have weight status within normal and to consume a healthy diet and engage in physical activity than toddlers with parents in a placebo (safety) intervention.

DETAILED DESCRIPTION:
Background:

Overweight is a serious public health problem which can begin in early childhood. Factors which contribute to overweight include: overfeeding, excessive intakes of fat and sugar; frequent sedentary activities (i.e. television watching).

Overweight, defined as a BMI > 95th percentile, in early childhood has reached epidemic proportions with 14% of 2-5 year olds overweight and 26.2% "at risk of overweight," defined as a BMI > 85th percentile (Ogden et al., 2006).

Dietary and physical activity patterns established early in life track over time, making the first few years of life an ideal time to help families establish healthy eating and physical activity behaviors and avoid overweight. This project works to identify techniques that could prevent overweight.

Purpose of Study:

The investigators are collaborating with the Anne Arundel County, MD Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) and the University of Maryland's Pediatric Ambulatory Center to implement strategies that will prevent overweight among toddlers. The project focuses on the dietary, physical activity, and growth patterns of WIC toddlers. The investigators are conducting a 3-cell randomized trial consisting of: 1) a maternal intervention focusing on healthy diet and physical activity patterns for mothers; 2) a toddler parenting intervention focusing on parenting, limit setting, and development strategies; and 3) an intervention on child safety. The interventions are implemented over 3 months, with 8 sessions.

The investigators hypothesize that altering maternal behavior will have a positive impact on the growth and development of the toddler by preventing behaviors that lead to overweight among children. The parenting intervention will improve parenting skills by offering information on proper approaches to feeding, discipline and educational play. The investigators will compare the growth patterns of toddlers whose mothers were randomized to the maternal and parenting interventions with those in the safety intervention. This study design allows us to examine the mechanisms linking the interventions to improvements in diet, physical activity, and growth.

In addition, the investigators will conduct the safety promotion intervention for the attention control group, considering the high risk of unintentional injuries among the toddlers from low-income families. The investigators also hypothesize that the safety promotion intervention will reduce the safety problems of the toddlers' homes. The underlying mechanisms will be examined, if there is a significant intervention effect.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 yrs old
* Has child between 12-32 months
* Child able to walk
* Birth weight of child at least 5lbs. 8oz.

Exclusion Criteria:

* Mom cannot be pregnant
* No known congenital problems or disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2006-04; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, PhD, Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - University of Maryland, School of Medicine, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Derived] Campbell KL, Wang Y, Kuhn AP, Black MM, Hager ER. An ecological momentary assessment study of physical activity behaviors among mothers of toddlers from low-income households. BMC Womens Health. 2021 Mar 22;21(1):120. doi: 10.1186/s12905-021-01243-2. PMID 33752659
- [Derived] Covington L, Armstrong B, Trude ACB, Black MM. Longitudinal Associations Among Diet Quality, Physical Activity and Sleep Onset Consistency With Body Mass Index z-Score Among Toddlers in Low-income Families. Ann Behav Med. 2021 Jun 28;55(7):653-664. doi: 10.1093/abm/kaaa100. PMID 33196078
- [Derived] Black MM, Hager ER, Wang Y, Hurley KM, Latta LW, Candelaria M, Caulfield LE. Toddler obesity prevention: A two-generation randomized attention-controlled trial. Matern Child Nutr. 2021 Jan;17(1):e13075. doi: 10.1111/mcn.13075. Epub 2020 Sep 4. PMID 32885909
- [Derived] Armstrong B, Covington LB, Hager ER, Black MM. Objective sleep and physical activity using 24-hour ankle-worn accelerometry among toddlers from low-income families. Sleep Health. 2019 Oct;5(5):459-465. doi: 10.1016/j.sleh.2019.04.005. Epub 2019 Jun 3. PMID 31171491
- [Derived] Wang Y, Gielen AC, Magder LS, Hager ER, Black MM. A randomised safety promotion intervention trial among low-income families with toddlers. Inj Prev. 2018 Feb;24(1):41-47. doi: 10.1136/injuryprev-2016-042178. Epub 2017 Apr 6. PMID 28385953
- See also: Study Website — https://www.medschool.umaryland.edu/growth/

RESULTS

PARTICIPANT FLOW:
Groups:
- Maternal Lifestyle (Physical Activity and Nutrition): A maternal lifestyle intervention focusing on healthy diet and physical activity patterns for mothers.
  Maternal Lifestyle (Physical Activity and Nutrition): At each session, mothers will identify a dietary goal for the next session (e.g., reduce soda intake). They will learn to track and evaluate their progress, setting new goals or modifying existing ones as necessary. Mothers will be given pedometers and shown how to keep a pedometer tracking chart. As with dietary choice, our objective is to have the mothers identify personal goals and strategies to achieve those goals, so they are more likely to continue to engage in physical activity after the intervention ends.
- Responsive Parenting: A responsive parenting intervention focusing on parenting, limit setting, and development strategies.
  Responsive Parenting: Behavior and Development Related to Diet and Physical Activity. The toddler parenting intervention will include modules on toddler behavior and development. We will devote sessions to topics involving parenting toddlers, limit setting, and child development.
Period: Overall Study
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Started | 94 | 92 | 91
Completed | 73 | 76 | 75
Not Completed | 21 | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety | Total
Number analyzed (Participants) | 94 | 92 | 91 | 277
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.17 (5.9) | 27.53 (6.5) | 28.16 (5.99) | 27.28 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 91 | 277
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 3 | 5
  Not Hispanic or Latino | 92 | 92 | 88 | 272
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 64 | 67 | 62 | 193
  White | 21 | 19 | 22 | 62
  More than one race | 7 | 6 | 5 | 18
  Unknown or Not Reported | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 94 | 92 | 91 | 277
Maternal age [Mean (Standard Deviation); unit: years] | 26.17 (5.9) | 27.53 (6.5) | 28.16 (5.99) | 27.28 (6.17)
Household Poverty Ratio [Count of Participants; unit: Participants] — Household poverty ratio was calculated based on the federal poverty threshold for the year the data were collected using mother-reported total family income and number of household members. We summed the number of families with poverty ratio below 1, indicating that the average income for the family size is below the official definition of poverty.
  Participants | 68 | 59 | 58 | 185
Maternal Education [Count of Participants; unit: Participants] — We calculated the number of mothers who had completed high school or the General Educational Development (GED) test.
  Participants | 74 | 75 | 75 | 224
Maternal Marital Status [Count of Participants; unit: Participants] — Count of the number of mothers who were married
  Participants | 24 | 25 | 29 | 78
Location (Urban/Semi-Urban) [Count of Participants; unit: Participants] — Families were recruited from 2 sites: urban and semi-urban. We counted the number of mothers from the urban site
  Participants | 56 | 58 | 53 | 167
Maternal BMI [Mean (Standard Deviation); unit: kg/m^2] — Weight and height are measured to calculate BMI (kg/m^2).
  kg/m^2 | 31.98 (9.48) | 31.90 (9.78) | 31.51 (9.24) | 31.80 (9.47)
Maternal dietary intake [Mean (Standard Deviation); unit: kcal/day] | 2281 (745) | 2214 (1053) | 2033 (738) | 2177 (859)
Maternal physical activity [Mean (Standard Deviation); unit: Minutes Mod/Vig Activity/Day] | 23.22 (18.07) | 26.14 (20.36) | 27.52 (17.82) | 25.54 (18.76)
Toddler age [Mean (Standard Deviation); unit: months] | 19.98 (5.55) | 20.22 (5.56) | 20.14 (5.46) | 20.11 (5.50)
Toddler sex [Count of Participants; unit: Participants]
  Females | 48 | 37 | 45 | 130
  Males | 46 | 55 | 46 | 147
Toddler race/ethnicity [Count of Participants; unit: Participants]
  Non-Hispanic African American | 64 | 67 | 62 | 193
  Non-Hispanic White | 21 | 19 | 22 | 62
  Hispanic | 2 | 0 | 3 | 5
  Mixed | 7 | 6 | 4 | 17
Toddler Body Mass Index (BMI) Z-score [Mean (Standard Deviation); unit: Body mass index z-scores] — Body Mass Index, kg/m^2, is calculated by measured weight and height. BMI z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. These scores are used to determine weight status (e.g., overweight, obese, etc.)
  Body mass index z-scores | 0.49 (1.10) | 0.51 (1.16) | 0.63 (1.14) | 0.54 (1.13)
Toddler dietary intake [Mean (Standard Deviation); unit: Total energy kcal/day] | 1282 (476) | 1297 (463) | 1262 (419) | 1281 (453)
Toddler physical activity [Mean (Standard Deviation); unit: Minutes Mod/Vig physical activity/day] | 45.45 (38.53) | 52.99 (35.87) | 64.62 (45.16) | 54.08 (40.43)

OUTCOME MEASURES:

1. Primary Outcome: Change of Body Mass Index (BMI) Z-score for Toddlers
Description: Measured weight and height for the toddlers, transferred to age and gender-specific body mass index (BMI) Z-score. The range of BMI z-score is usually between -5 and +5. BMI z-score lower than -1.645 is defined as underweight. The BMI z-score from -1.645 to 1.036 is normal weight and BMI z-score greater or equal to 1.645 is obese.
Time Frame: Baseline to 12-month Follow-up
Population: Toddlers in low-income families, defined as WIC-eligible (income < 185% of poverty index). WIC=Special Supplementary Program for Women, Infants, and Children.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
z-score
  Toddlers BMI z-score at baseline | 0.49 (0.12) | 0.50 (0.12) | 0.62 (0.12)
  Toddler BMI z-score12-month follow-up | 0.52 (0.12) | 0.61 (0.12) | 0.57 (0.12)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; H0: There are no differences between the maternal lifestyle and child safety groups in the change in BMI z-score over time. Mixed models included the interaction between time and intervention, accounting for clustering of the repeated measures within each individual; Test type: Equivalence — If the 95% confidence interval of the difference in the change over time does not include 0, it means that there is a significant difference in the change over time between the two groups; p = 0.555, Mixed Models Analysis — The alpha for statistical significance is set at 0.05; Slope = 0.07, 95% CI 2-sided [-0.17 to 0.31], Standard Error of Mean 0.12 — This is to compare change in maternal lifestyle group to child safety group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; Test type: Equivalence — 95% CI; p = 0.200, Mixed Models Analysis — Two-side test; Slope = 0.16, 95% CI 2-sided [-0.08 to 0.39], Standard Error of Mean 0.12 — This is to compare the Responsive Parenting to the safety intervention group

2. Primary Outcome: Change in Body Mass Index (BMI) Score Among Mothers
Description: Change body mass index (BMI, kg/m^2, calculated by measured weight and height) from baseline to 12-month follow-up. The BMI ranges usually ranges from 0-50 with higher score indicating higher weight regarding the height. Scores above 25 are considered overweight and scores above 30 are considered obese.
Time Frame: Baseline to 12 month Follow-up
Population: Mothers of toddlers participating in study, low-income, defined as WIC-eligible.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
kg/m^2
  Maternal BMI at baseline | 31.98 (0.98) | 31.90 (0.99) | 31.51 (0.99)
  Maternal BMI at 12-month follow-up | 32.22 (0.99) | 32.21 (0.99) | 31.85 (1.00)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; H0: There is no difference between maternal lifestyle and child safety groups in the change of BMI over time; Test type: Equivalence — 95% confidence interval (CI) was estimated. If the 95% CI does not include 0, it means there is significant difference in the change over time between the two groups; p = 0.739, Mixed Models Analysis — The alpha for statistical significance is set at 0.05; Slope = -0.11, 95% CI 2-sided [-0.74 to 0.52], Standard Error of Mean 0.32 — This is to compare maternal lifestyle to child safety group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; H0: There are no differences in the change over time between responsive parenting and child safety groups; Test type: Equivalence — The 95% CI was estimated. If it does not include 0, it means that there is a statistically significant difference in the change over time between the two groups; p = 0.904, Mixed Models Analysis — The alpha for statistical significance was set at 0.05; Slope = -0.04, 95% CI 2-sided [-0.66 to 0.59], Standard Error of Mean 0.32 — This is to compare the responsive parenting group to the child safety group

3. Secondary Outcome: Change of Diet Quality for Toddlers
Description: Healthy Eating Index 2015 (HEI 2015) based on 24-hr diet recall. The range is 0-100, with higher scores representing better diet quality.
Time Frame: Baseline to 12-month Follow-up
Population: Change in HEI 2015 score for toddlers from baseline to 12 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
units on a scale
  Toddler HEI total at baseline | 52.44 (1.18) | 54.58 (1.20) | 55.1 (1.19)
  Toddler HEI total at 12-month follow-up | 52.84 (1.38) | 52.49 (1.36) | 52.19 (1.35)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; H0 is that there is no difference between maternal lifestyle and child safety groups in the change of HEI 2015 score over time; Test type: Equivalence — The 95% confidence interval (CI) for the difference in the change over time was estimated. If it does not include 0, it indicates significant difference in the change over time; p = 0.168, Mixed Models Analysis — Alpha is set at 0.05; Slope = 3.31, 95% CI 2-sided [-1.4 to 8.02], Standard Error of Mean 2.40
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; H0 is that there is no difference between the responsive parenting and child safety groups in the change of HEI score over time; Test type: Equivalence — 95% CI was estimated. If it does not include 0, it indicates that there is a significant difference in the change between the two groups; p = 0.733, Mixed Models Analysis; Slope = 0.82, 95% CI 2-sided [-3.88 to 5.52], Standard Error of Mean 2.39 — This is to compare the responsive feeding group to child safety group

4. Secondary Outcome: Change of Diet Quality for Mothers
Description: Healthy Eating Index (HEI 15) is calculated based on 24 hour diet recall. Scores range from 0-100, with higher scores optimal
Time Frame: Baseline to 12-month Follow-up
Population: Mothers of toddlers
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
score on a scale
  Baseline HEI 2015 | 46.88 (1.32) | 48.71 (1.35) | 48.52 (1.34)
  12-month HEI 2015 | 48.39 (1.52) | 46.90 (1.53) | 46.74 (1.57)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; Null hypothesis is that there are no differences between the two groups regarding the change of HEI 2015 score over time; Test type: Equivalence — The 95% CI was estimated. If it does not include 0, it indicates that there is significant difference in the change over time between the two groups; p = 0.186, Mixed Models Analysis — Alpha is set at 0.05; Slope = 3.30, 95% CI 2-sided [-1.6 to 8.2], Standard Error of Mean 2.49 — This is to compare the maternal lifestyle group to the child safety group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; H0 is there is no difference in the change of maternal HEI score over time between the two groups; Test type: Equivalence — 95% CI for the difference in change over time was estimated. If it does not include 0, it indicates that there is significant difference between the two groups; p = 0.990, Mixed Models Analysis — Alpha is set to 0.05; Slope = -0.03, 95% CI 2-sided [-4.97 to 4.91], Standard Error of Mean 2.51 — This is to compare the responsive parenting group to child safety group

5. Secondary Outcome: Change of Child Physical Activity
Description: Physical activity is measured by wearing an accelerometer for 7 days. Using standards for toddlers, we count the number of minutes in moderate-vigorous physical activity (MVPA) per day, and averaged over the number of days measured, higher scores mean more physical activity.
Time Frame: Baseline to 12-month Follow-up
Population: Toddlers who participated in the trial, from low-income families, defined as WIC-eligible
Measure: Mean (Standard Error); unit: minutes per day
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
minutes per day
  Toddler MVPA at baseline | 44.56 (4.92) | 52.39 (4.98) | 64.18 (5.11)
  Toddler MVPA at 12-month follow | 73.10 (7.37) | 71.05 (7.13) | 69.05 (7.14)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; Null hypothesis is there were no differences in the change over time for toddler MVPA across the two groups; Test type: Equivalence — A 95% CI was estimated. If it does not include 0, it indicates significant difference in change over time between the two groups; p = 0.034, Mixed Models Analysis — Alpha is set at 0.05; Slope = 23.67, 95% CI 2-sided [1.88 to 45.46], Standard Error of Mean 11.03 — This is for maternal lifestyle group compared to safety control group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; Test type: Equivalence — H0 is that there is no difference between the change of MVPA over time between the two groups; p = 0.216, Mixed Models Analysis; Slope = 13.52, 95% CI 2-sided [-7.98 to 35.03], Standard Error of Mean 10.89 — This is to compare the responsive parenting group to child safety group

6. Secondary Outcome: Change of Maternal Physical Activity
Description: Physical activity is measured by wearing an accelerometer for 7 days. Using standards for adults, we count the number of minutes in moderate-vigorous physical activity (MVPA) per day, and averaged over the number of days measured, higher scores mean more physical activity.
Time Frame: Baseline-12 month follow up
Population: Change in the number of steps per day from baseline to 12-month follow-up in MVPA
Measure: Mean (Standard Error); unit: minutes per day
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
minutes per day
  Maternal MVPA at baseline | 23.10 (2.06) | 26.11 (2.17) | 27.76 (2.17)
  Maternal MVPA at 12-month follow | 27.41 (3.07) | 20.42 (3.21) | 21.09 (3.22)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; H0 is that there is no difference in the change of maternal MVPA over time between the two groups; Test type: Equivalence — The 95% CI for the difference in the change between the two groups was estimated. If it does not include 0, it indicates that there is a significant difference by group in the change; p = 0.024, Mixed Models Analysis; Slope = 10.97, 95% CI 2-sided [1.46 to 20.48], Standard Error of Mean 4.82 — This is to compare the maternal lifestyle group to the child safety group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; H0 is that there is no significant difference in the change of maternal MVPA between the two groups; Test type: Equivalence — The 95% CI was estimated. If it does not include 0, it indicates that there is a significant difference by group in the difference; p = 0.804, Mixed Models Analysis; Slope = 0.98, 95% CI 2-sided [-8.76 to 10.72], Standard Error of Mean 4.94 — This is to compare responsive parenting group to child safety group

7. Secondary Outcome: Feeding Style
Description: The Emotional Availability Scales (EAS) include 4 maternal scales (sensitivity, structuring, non-intrusiveness, and non-hostile) and 2 child scales (responsiveness and involvement), each rated on 7-point Likert scales, with high scores optimal. The maternal and child sub-scale scores were averaged for a total mealtime interaction score. The total score ranges from 1-7. Coders were trained until they demonstrated inter-rater reliability >0.80 based on intraclass correlation coefficients with 10 observations from the scale creator and 10 observations with the faculty coordinator. Inter-rater reliability was reviewed through weekly reliability checks.
Time Frame: Baseline to 12 month Follow-up
Population: Change in Emotional Availability Scale scores from baseline to 12-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
Number analyzed (Participants) | 94 | 92 | 91
score on a scale
  Maternal feeding style at baseline | 4.69 (0.11) | 4.42 (0.11) | 4.71 (0.12)
  Maternal feeding style at 12-month | 5.07 (0.14) | 5.19 (0.14) | 5.46 (0.13)
Statistical Analysis 1: Comparison: Maternal Lifestyle (Physical Activity and Nutrition) vs Child Safety; The 95% CI was estimated. If it does not include 0, it indicates that there is a significant difference by group in the difference; Test type: Equivalence — [test comment as in outcome 6, analysis 2]; p = 0.056, Mixed Models Analysis — Alpha is set at 0.05 for statistical significance; Slope = -0.36, 95% CI 2-sided [-0.78 to 0.06], Standard Error of Mean 0.21 — This is to compare maternal lifestyle group to the child safety group
Statistical Analysis 2: Comparison: Responsive Parenting vs Child Safety; [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — Alpha is set at 0.05 to indicate statistical significance; p = 0.896, Mixed Models Analysis; Slope = 0.03, 95% CI 2-sided [-0.39 to 0.45], Standard Error of Mean 0.21 — This is to compare responsive parenting group to child safety group

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the time period that participants were actively participating in the study and assessments (e.g., 12 months for each participant or until the final assessment was completed).
Description: Data Safety Monitoring Committee reviewed records and interviewed project coordinator.
Arm/Group | Maternal Lifestyle (Physical Activity and Nutrition) | Responsive Parenting | Child Safety
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 0/94 | 0/92 | 0/91

LIMITATIONS AND CAVEATS:
Data analysis was delayed due to extended period of time for coding the mother-toddler interaction data, related to personnel and funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No